CLINICAL TRIAL: NCT00651339
Title: The Effect of Botox Injection on Postural Stability of Cerebral Palsy (CP) Children
Status: Terminated | Type: Observational
Why Stopped: recruiting or enrolling participants has halted prematurely and will not resume
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Itshak Melzer PhD, PT, Ben-Gurion University of the Negev
Other Study IDs: sor465708ctil
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2008-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Balance; Gait
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A
  Interventions: Drug: botox

INTERVENTIONS:
Drug: botox — botox injection

SUMMARY:
Children suffer from Cerebral Palsy that willing to participate in the study will be tested with well-established measuring techniques of Balance control using force plate before 2 month after BOTOX injection in the movement and Rehabilitation Laboratory at BGU. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). Each of the Times (before 3 month and 6 month after the THA) in two task conditions (eyes closed and eyes close conditions). Participants will be required to stand on the platform 5 times for 30 s For each trial, they will be instructed to sway as little as possible. In addition Gait analysis will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* BOTOX injection

Exclusion Criteria:

* Not able to stand independently 60 seconds
* Not able to walk independently

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 children suffer from Cerbral Palsy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
SDF parameters | before and 2 months after the BOTOX injection

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel